CLINICAL TRIAL: NCT03910777
Title: Usefulness of Early Warning Systems in Detecting Early Clinical Deterioration After Intensive Care Discharge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, ILKE KUPELI, assist. prof., Erzincan University
Other Study IDs: EBYU 2
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Early Clinical Deterioration; Early Warning Score
MeSH Terms: conditions — Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Early Warning Score — National early warning score (NEWS) is another early warning scoring system recommended by the Royal College of Physicians in London to detect early clinical deterioration in hospitalized patients

SUMMARY:
The VitalPac Early Warning Score (VIEWS) scoring system, developed by Prytherch et al., Is an early warning system that aims to predict the first 24-hour mortality in emergency patients.

National early warning score (NEWS) is another early warning scoring system recommended by the Royal College of Physicians in London to detect early clinical deterioration in hospitalized patients.

The aim of this study was to determine the early clinical deterioration after ICU and hence the rate of admission to intensive care and to evaluate whether these two scoring systems can be used to determine early clinical deterioration in intensive care early discharge.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years,
* discharged from the ICU and returned within 24 hours

Exclusion Criteria:

* under 18 years old, postoperative patients, pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 390 patients who were discharged from the intensive care unit over the age of 18 and who were taken back within 24 hours will be included.
Sampling Method: Non-Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of patients recovered due to early clinical deterioration within the first 24 hours after ICU discharge | six month
  The aim of this study is to determine the early clinical deterioration in the first 24 hours after ICU discharge and therefore the rate of admission to ICU.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Uppanisakorn S, Bhurayanontachai R, Boonyarat J, Kaewpradit J. National Early Warning Score (NEWS) at ICU discharge can predict early clinical deterioration after ICU transfer. J Crit Care. 2018 Feb;43:225-229. doi: 10.1016/j.jcrc.2017.09.008. Epub 2017 Sep 13. PMID 28926736
- [Result] Cardoso FS, Karvellas CJ, Kneteman NM, Meeberg G, Fidalgo P, Bagshaw SM. Respiratory rate at intensive care unit discharge after liver transplant is an independent risk factor for intensive care unit readmission within the same hospital stay: a nested case-control study. J Crit Care. 2014 Oct;29(5):791-6. doi: 10.1016/j.jcrc.2014.03.038. Epub 2014 Apr 24. PMID 24857401